CLINICAL TRIAL: NCT06369571
Title: Improving Cardiovascular Health Risks in Adults With Epilepsy on a Modified Atkins Diet
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00439268
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy; Dyslipidemia
Keywords: Modified Atkins Diet; Ketogenic Diet; Cholesterol
MeSH Terms: conditions — Epilepsy; Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Statin (Active Comparator): Participants will receive 10mg of atorvastatin daily for 12 weeks
  Interventions: Drug: Atorvastatin 10mg
- Modified Atkins diet (MAD) Modification (Experimental): Participants will be instructed on how to change their modified Atkins diet for 12 weeks. They will replace 10% of daily dietary energy from saturated fat with poly-unsaturated fat.
  Interventions: Other: Modification of dietary fat composition

INTERVENTIONS:
Drug: Atorvastatin 10mg — Atorvastatin 10mg daily by mouth
  Other Names: Lipitor
  Arms: Statin
Other: Modification of dietary fat composition — Replace 10% of saturated fat intake with polyunsaturated fat
  Arms: Modified Atkins diet (MAD) Modification

SUMMARY:
Ketogenic diet therapies (KDTs) emphasize high fat and very low carbohydrate intake and help to control seizures in adults who fail to respond to medications. However, KDT use can lead to increased cholesterol levels in some adults with epilepsy (AWE). Treatments that can reverse elevations in cholesterol observed with long-term KDT use without compromising diet adherence and seizure control are needed. The proposed study will explore the feasibility and safety of diet modification and statin use to lower cholesterol in this population. Study findings will help guide doctors utilizing KDTs in adults with epilepsy on how to approach managing elevations in cholesterol.

DETAILED DESCRIPTION:
The scientific premise of this proposal is that established or long-term (≥ 12 months) Modified Atkins diet (MAD) use in AWE influences atherosclerotic cardiovascular disease (ASCVD) risk and can be modified to reduce dyslipidemia when observed. Hence, the overarching goals of this proposal are to explore the safety and feasibility of dyslipidemia management strategies to reduce ASCVD risk in AWE on MAD without increasing seizure risk. This study will collect data before and after randomly assigned interventions to reduce LDL in AWE on long-term MAD recruited from patients receiving clinical care in the Johns Hopkins Adult Epilepsy Diet Center.

AWE with dyslipidemia on long-term MAD will be randomized 1:1 to either MAD modification (10% reduction of dietary energy from saturated fat, replaced with poly-unsaturated fat ) or moderate-intensity statin use (atorvastatin 10mg) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Modified Atkins Diet use ≥ 12 months
2. Dyslipidemia based on American College of Cardiology/American Heart Association guidelines (i.e., LDL ≥190 mg/dL, 10-year ASCVD risk ≥5% with risk enhancers, etc.)
3. 18 years of age or older
4. Body mass index (BMI) > 18.5
5. Stable anti-seizure medication regimen for > 1 month.

Exclusion Criteria:

1. < 18 years of age
2. Body mass index (BMI) < 18.5
3. Changes in anti-seizure medication regimen < 1 month prior to participation
4. Known ASCVD (history of acute coronary syndrome, myocardial infarction, angina, stroke, transient ischemic attack, or peripheral artery disease)
5. Current statin medication use
6. Prior serious adverse response to atorvastatin or other statin medications
7. Uncorrected carnitine deficiency
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Diet adherence as assessed by 3 day food records | 12 weeks
  Diet adherence will be based on the ability to achieve 10% reduction in dietary energy from saturated fat assessed from 3-day food records, the gold standard for diet intake assessments.
Statin Adherence | 12 weeks
  Statin adherence will be determined based on pills returned at study completion, with participants labeled adherent if 80% or more of pills were consumed.
LDL Change | 12 weeks
  12-week % LDL change from baseline within arms and between arms
Change in weekly seizure frequency | 12 weeks
  12-week difference in weekly seizure frequency from baseline
Seizure severity questionnaire score | 12 weeks
  12-week difference in seizure severity questionnaire (SSQ) score (score 1-7, with higher score indicating more severe seizures)

SECONDARY OUTCOMES:
Frequency of adverse events | 12 weeks
  Frequency of adverse events
Blood ketone change | 12 weeks
  12-week difference in serum beta-hydroxybutyrate level from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tanya J McDonald, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No